CLINICAL TRIAL: NCT04048642
Title: Effects of a Plant-Based Diet on Insulin Requirements and Obesity Markers in Obese Adults With T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Thomas M Campbell, Assistant Professor of Family Medicine, University of Rochester
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003764
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Resistance; Obesity; Nutritional and Metabolic Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Obesity; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DASH diet; plant-based diet; DASH diet (Experimental): Food is provided: 7 days of an ad libitum DASH diet, followed immediately by 7 days of an ad libitum whole food, plant based diet, followed immediately by 7 days of an ad libitum DASH diet again.
  Interventions: Behavioral: DASH; Behavioral: Whole-Food, Plant-Based

INTERVENTIONS:
Behavioral: DASH — 7 days of a DASH diet
Behavioral: Whole-Food, Plant-Based — 7 days of a WFPB diet

SUMMARY:
This is a crossover study utilizing a Dietary Approaches to Stop Hypertension (DASH) diet and a whole-food, plant-based diet among subjects with type 2 diabetes who require insulin. Outcomes are short-term changes in insulin requirements and changes in various biomarkers.

DETAILED DESCRIPTION:
This is a single center, prospective, non-randomized crossover study. The aim of the study is to perform a comprehensive evaluation of factors that may contribute to improvements in glycemic control in obese patients with type 2 diabetes during a plant-based dietary intervention. The primary end point will be the change in total daily insulin requirements during the plant-based dietary intervention period compared against a Dietary Approaches to Stop Hypertension (DASH) diet. Evaluation of insulin requirements will be carried out in three phases of this study: pre-intervention (Phase 1), intervention (Phase 2), and post-intervention (Phase 3). Each phase is 7 days. In addition, investigators plan to evaluate the effects of a plant-based diet on glucose homeostasis by estimating the insulin sensitivity index and beta cell function using weekly sampled oral glucose tolerance tests (oGTT) and will explore if these effects correlate with changes in urinary glucose excretion by using weekly sampled urinary tests. Investigators will also be assessing changes in obesity-related inflammatory biomarkers, stress biomarkers and metabolic markers during the three phases of the study. Lastly, given the current technological advantages in the field of diabetes monitoring, investigators plan to monitor the glycemic excursion curve using a continuous glucose monitor during the complete study.

ELIGIBILITY:
Inclusion Criteria:

* Adults (older than 18 years old) of both genders, of all races and ethnicities.
* Pre-existing diagnosis of Type 2 Diabetes Mellitus, as documented in medical records on basal with or without mealtime bolus insulin with no change to total of basal insulin and nutritional baseline insulin dosing > 10% in the 1 month prior to consent and no changes to non-insulin antihyperglycemic medications in the 3 months prior to consent
* If on a GLP-1 analog, on a stable dose for at least 3 months prior to the study enrollment
* If on an SGLT2 inhibitor, on a stable dose for at least 3 months prior to the study enrollment
* BMI of 27 kg/m2 or greater
* Most recent HbA1c (within 6 months prior to consent) between 6.5% and 9.5%
* Fluent in the English language (education about each diet will be in English)
* Willingness and ability to participate in study protocol.
* Agreeable to give informed consent.

Exclusion Criteria:

* Diagnosis of T1DM or type 1.5 diabetes mellitus
* History of liver cirrhosis
* Impaired renal function (GFR < 45 ml/min) within 6 months prior to consent
* History of hyperkalemia (potassium > 5.4 meq/L) within 6 months prior to consent
* Use of an insulin pump or expected to start during the study period
* Use of warfarin (Coumadin)
* Use of daily aspirin 500 mg or more or expected to start during the study period
* Use of daily Vitamin C of 1,000 mg or more, unless willing to stop taking 1 week prior to baseline visit and for duration of study
* Use of antipsychotics or systemic steroids within 3 months prior to consent
* Use of any of the following weight-lowering pharmacotherapy within 3 months prior to consent: phentermine, orlistat, lorcaserin, phentermine/topiramate, bupropion/naloxone
* The use of insulin secretagogues including sulfonylureas and glinides within 3 months prior to consent as this may increase the risk of hypoglycemia and alter assessment of daily insulin requirements during the study
* The use of illicit drugs, defined as active use or use within 3 months prior to consent.
* Engage in high risk alcohol use (defined as more than 4 drinks on any day or more than 14 drinks per week in men and more than 3 drinks on any day or 7 drinks per week in women).
* Individuals who are pregnant or breastfeeding or intend to become pregnant during the duration of the study
* Individuals who are following a vegetarian or vegan diet at the time of consent
* Food allergies or intolerances that will interfere with diet adherence
* Lack of access to a full-size refrigerator (required for storage of 3-4 days of prepared study meals)
* Active malabsorption disorder, including uncontrolled symptomatic inflammatory bowel disease, or bariatric surgery in the past 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Change in total daily insulin requirements | 7 Days

SECONDARY OUTCOMES:
Changes in glucose excursion curve | 7 days
Changes in serum leptin | 7 days
Changes in serum adiponectin | 7 days
Changes in serum C-peptide levels | 7 days
Changes in serum insulin levels | 7 days
Change in lipid panel | 7 days
Change in hsCRP | 7 days
Change in IL-6 | 7 days
Change in IL-18 | 7 days
Change in TNF-a | 7 days
Change in urinary catecholamines | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Jonven Attia, MD, Principal Investigator — University of Rochester; Thomas M Campbell, MD, Principal Investigator — University of Rochester
Locations (1):
- UR Medicine/Highland Hospital Nutrition in Medicine Research Center, Webster, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Campbell EK, Taillie L, Blanchard LM, Wixom N, Harrington DK, Peterson DR, Wittlin SD, Campbell TM. Post hoc analysis of food costs associated with Dietary Approaches to Stop Hypertension diet, whole food, plant-based diet, and typical baseline diet of individuals with insulin-treated type 2 diabetes mellitus in a nonrandomized crossover trial with meals provided. Am J Clin Nutr. 2024 Mar;119(3):769-778. doi: 10.1016/j.ajcnut.2023.12.023. Epub 2023 Dec 30. PMID 38160802